CLINICAL TRIAL: NCT02845076
Title: Weaning From Noninvasive Ventilation
Acronym: WEANIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: University of Bologna (Other); Marmara University (Other); Istanbul Sureyyapasa Chest Diseases and Chest Surgery Training and Research Hospital (Other); Dokuz Eylul University (Other); Cukurova University (Other); Ospedale San Donato (Other); University of Milan (Other)
Responsible Party: Principal Investigator, Aylin Ozsancak Ugurlu, MD, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BaskentU
Record Dates: First submitted 2016-03-28; First posted 2016-07-27 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Hypercapnic Respiratory Failure; Weaning Failure; Noninvasive Ventilation
Keywords: Noninvasive ventilation; Respiratory insufficiency; Hypercapnia; ventilator weaning
MeSH Terms: conditions — Respiratory Insufficiency; Hypercapnia | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Decrease in duration (Active Comparator): Weaning will be started with the liberation of patient from NIV during day-time and then nighttime support will be gradually reduced. From day 2 the daytime NIV will be gradually decreased in steps of at least 2 hours/day at the attending discretion. At day 2, nighttime discontinuation will be considered. When a patient reaches without the presence of any reinstitution criteria, the duration of NIV use as 4 hours per 16 hours during daytime, it will be liberated definitively from NIV.
  Interventions: Other: Protocol for weaning of noninvasive ventilation
- Decrease in pressure and duration (Active Comparator): Weaning will be started with the liberation of patient from NIV during day-time and then nighttime support will be gradually reduced. The level of pressure support will be decreased by 2-4 cmH2O per 4 hours during daytime in patients with good tolerance, with no change at night time. From day 2 the daytime NIV will be gradually decreased in steps of at least 2 hours/day at the attending discretion. At day 2, nighttime discontinuation will be considered, based on the vitals and ABGs recorded at 8 pm (see above), with gradual decrease of at least 2 hrs/night. When a patient reaches without the presence of any reinstitution criteria, the level of PS of 8 cmH20, it will be liberated definitively from NIV.
  Interventions: Other: Protocol for weaning of noninvasive ventilation
- Abrupt discontinuation of NIV (Active Comparator): Patients will be disconnected from NIV and oxygenated with a nasal cannula. Oxygen flow will be limited to a maximum of 5L/min.
  Interventions: Other: Protocol for weaning of noninvasive ventilation

INTERVENTIONS:
Other: Protocol for weaning of noninvasive ventilation — 3 protocols for weaning of noninvasive ventilation will be compared

SUMMARY:
Noninvasive ventilation (NIV) weaning strategies differ considerably from one another. These strategies have yet not been compared to each other. Therefore, the investigators planned to perform a prospective, randomized, pilot study involving hypercapnic acute respiratory failure patients ready to be weaned off from NIV. The investigators are going to compare the success rate of NIV weaning and the duration of NIV after randomization between 3 NIV weaning methods: gradual decrease in duration of NIV or level of ventilator support, and abrupt discontinuation of NIV.

ELIGIBILITY:
Inclusion Criteria:

Patients will be screened by the physician 24 hours (±6 hours) after initiation of NIV treatment if:

* Age ≥18 years old
* Hypercapnic ARF ( baseline pH<7.35, paCO2>45 mmHg, BORG>4)
* Breathing frequency< 25 bpm under NIV
* pH >7.35 under NIV
* 10% or more decrease from baseline PaCO2 under NIV
* Kelly ≤ 2 under NIV (Alert. Follows simple/3 step complex commands)
* PaO2 between 60 and 70 mmHg under NIV
* No need for sedation
* Systolic blood pressure 90-180 mmHg without vasopressors
* Body temperature 36-38°C
* Heart rate 50-120 bpm

The patient will be enrolled to the study and will be randomized to one of the NIV weaning protocols, if passes daily weaning criteria listed below after 1 hour of spontaneous breathing (with supplementary oxygen),

* Respiratory rate 8-30 bpm
* Systolic blood pressure 90-180 mmHg without vasopressors
* Body temperature 36-38°C
* Heart rate 50-120 bpm
* Neurologic score of Kelly ≤2 (Alert. Follows simple/ 3-step complex commands),
* SaO2 ≥88-92% with a FiO2≤40%.
* pH≥7.35
* Absence of severe dyspnea (BORG>4).

Exclusion Criteria:

* Age <18 years old
* NIV use at home for chronic respiratory failure
* CPAP use for acute respiratory failure
* NIV use as palliative treatment
* Severe heart failure with cardiac index ≤ 2 L/min/m2
* Severe hepatic failure with bilirubin ≥ 34.2µmol/L
* Severe renal failure with creatinine ≥ 220 µmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
The comparison of total duration of NIV after randomization | up to 10 days
  The patients will be considered as 'weaning failure' if:
  * The participant will meet the NIV reinstitution or intubation criteria during the weaning phase or within the first 5 days of NIV discontinuation
  * Weaning from NIV was not possible If the failing patient stabilizes afterwards and passes the screening and weaning criteria, the patient will be weaned again with the same protocol. If the patient fails weaning trials 3 times, then the patient will not be re-considered for further enrollment.

SECONDARY OUTCOMES:
Rate of NIV re-institution | 10 days of NIV discontinuation
NIV weaning success rates | 10 days of NIV discontinuation
Duration of ICU stay | up to 24 weeks
Rates of intubation | first 5 days of NIV discontinuation
In-hospital mortality | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nava, Study Chair — Bologna University; Begum Ergan, Study Director — Dokuz Eylul University; Sait Karakurt, Principal Investigator — Marmara University; Ezgi Ozyılmaz, Principal Investigator — Cukurova University; Raffaele Scala, Principal Investigator — San Donato Hospital; Fabiano Di Marco, Principal Investigator — Milan University; Zuhal Karakurt, Principal Investigator — Sureyyapasa Center for Chest Diseases and Thoracic Surgery Training and Investiagation Hospital
Locations (8):
- Italy (3):
  - San Donato Hospital, Arezzo
  - Bologna University, Bologna
  - Milan University, Milan
- Turkey (Türkiye) (5):
  - Cukurova University, Adana
  - Sureyyapasa Center for Chest Diseases and Thoracic Surgery Training and Investiagation Hospital, Istanbul
  - Baskent University, Istanbul
  - Marmara University, Istanbul
  - Dokuz Eylul University, Izmir

IPD SHARING:
Plan to Share IPD: Undecided